CLINICAL TRIAL: NCT03181724
Title: A Randomized Trial Measuring the Effect of Review of a Decision Aid Prior to the Appointment on Decisional Conflict Compared to Usual Care in the Treatment of Trapeziometacarpal (TMC) Arthritis
Brief Title: The Effect of Review of a Decision Aid Prior to the Appointment on Decisional Conflict Compared to Usual Care in the Treatment of Trapeziometacarpal (TMC) Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015P002550
Record Dates: First submitted 2017-06-02; First posted 2017-06-09 (Actual); Results first posted 2019-01-09 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Trapeziometacarpal Arthritis
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decision Aid (Active Comparator): Cohort that will receive a decision aid.
  Interventions: Behavioral: Decision Aid
- No Decision Aid (control) (No Intervention): One cohort will not receive the decision aid, and instead will receive only a brochure as standard treatment.

INTERVENTIONS:
Behavioral: Decision Aid — Cohort I will be managed with a decision aid (henceforth "DA"), and Cohort II will be managed without one. The patients in Cohort I will receive the DA, which they can complete in a separate room and take home. The decision aids include information on the disease/condition, treatment options, benefits, risks, scientific uncertainties, and probabilities of potential outcomes tailored to the patient's health risks factors. Additionally, it includes values clarifications such as describing outcomes in functional terms, asking patients to consider which benefits and risks matter most to them, and guidance in the steps of decision making and discussing their decision with family/friends. It is interactive and dynamic, helping patients clarify their preferences and come to a decision that feels best to them.
  Arms: Decision Aid

SUMMARY:
The investigators plan a prospective randomized controlled study that compares whether the use of a decision aid results in different scores on variables reflective of the decision-making process, behavior, health outcomes, communication, and healthcare system.

DETAILED DESCRIPTION:
Decision aids (shared decision making tools-websites, videos, or pamphlets) are interventions to prepare patients to make more informed decisions and satisfying decisions that match their preferences and values. With greater understanding of the risks and benefits of the treatment options patients may make a more informed choice.

Decision aids - delivered online, on paper, or on video - increase patient participation in the decision-making process,1 and can result in a decrease in discretionary surgery for knee osteoarthritis, herniated disk, and benign prostatic hypertrophy.2-4 They also reduce decisional conflict. Relatively few studies have investigated the influence of decision aids in orthopedic or hand surgery. Decision aids might affect decisional conflict, satisfaction, and outcomes in hand surgery where many treatments are discretionary and address quality of life.

Utilizing the Ottawa Decision Support Framework- an evidence-based, practical theory used to guide the development of decision aids - and the International Patient Decision Aid Standards criteria the investigators developed a decision aid for trapeziometacarpal arthritis.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* English-speaking
* Diagnosis of trapeziometacarpal (TMC) arthritis

Exclusion Criteria:

* Prior surgical intervention for trapeziometacarpal (TMC) arthritis
* Previously accessed or used the online TMC arthritis Decision Aid (DA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- [Background] Deyo RA, Cherkin DC, Weinstein J, Howe J, Ciol M, Mulley AG Jr. Involving patients in clinical decisions: impact of an interactive video program on use of back surgery. Med Care. 2000 Sep;38(9):959-69. doi: 10.1097/00005650-200009000-00009. PMID 10982117
- [Background] Jayadev C, Khan T, Coulter A, Beard DJ, Price AJ. Patient decision aids in knee replacement surgery. Knee. 2012 Dec;19(6):746-50. doi: 10.1016/j.knee.2012.02.001. Epub 2012 Mar 2. PMID 22386538
- [Background] Murray E, Davis H, Tai SS, Coulter A, Gray A, Haines A. Randomised controlled trial of an interactive multimedia decision aid on benign prostatic hypertrophy in primary care. BMJ. 2001 Sep 1;323(7311):493-6. doi: 10.1136/bmj.323.7311.493. PMID 11532845

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Decision Aid | No Decision Aid (Control)
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid | No Decision Aid (Control) | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.8) | 65.1 (9.8) | 63.7 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 65
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 43 | 40 | 83
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 45 | 90
Stage of Arthritis [Count of Participants; unit: Participants] — Determined radiographically using Eaton I-IV
  Participants
    Eaton stage I | 10 | 8 | 18
    Eaton stage II | 25 | 22 | 47
    Eaton stage III | 8 | 13 | 21
    Eaton stage IV | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Decision Conflict Scale (DCS)
Description: This scale measures patients' perception of uncertainty in making health-related decisions and consists of 3 subscales: (1) uncertainty choosing between different options, (2) modifiable factors contributing to this uncertainty-feeling uninformed, unclear about personal values, and feeling unsupported, and (3) perceived effectiveness of the decision-making an informed and values-based choice and expressing satisfaction with the decision. We used the validated statement format Decisional Conflict Scale, consisting of 16 items with 5 response options. Total scores range from 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Time Frame: Day 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Decision Aid | No Decision Aid (Control)
Number analyzed (Participants) | 45 | 45
units on a scale | 9.3 (1.9) | 17 (2)

2. Secondary Outcome: QuickDASH (Disabilities of the Arm, Shoulder and Hand) Questionnaire
Description: The short form of the Disabilities of Arm Shoulder and Hand to assess upper extremity disability. The scale range is from 0-100, where 0 is no difficulty performing tasks and 100 is the most difficulty or unable to complete any tasks.
Time Frame: Day 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Decision Aid | No Decision Aid (Control)
Number analyzed (Participants) | 45 | 45
units on a scale | 5.3 (.34) | 5.6 (.35)

3. Secondary Outcome: Patient Health Questionnaire-2 (PHQ-2)
Description: The PHQ-2 screens for depressive mood over the past 2 weeks. The score ranges from 0-6, where 0 is not at all depressed and 6 is major depression.
Time Frame: Day 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Decision Aid | No Decision Aid (Control)
Number analyzed (Participants) | 45 | 45
units on a scale | 0.44 (0.18) | 0.98 (0.25)

4. Secondary Outcome: Consultation and Relational Empathy (CARE) Measure
Description: The CARE measure is a 10-item questionnaire capturing patient perception of the physician's empathetic understanding under the office visit. Each item is rated on a 5-point Likert scale, yielding a total score from 0-50. A higher score indicates greater empathy.
Time Frame: Day 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Decision Aid | No Decision Aid (Control)
Number analyzed (Participants) | 45 | 45
units on a scale | 47 (0.84) | 45 (1.0)

5. Secondary Outcome: 11-point Ordinal Satisfaction Scale
Description: The patient satisfaction scale measures how satisfied a patient is with their treatment for their thumb arthritis. Patients score satisfaction on a scale of 0 to 10, where 0 is not satisfied and 10 is extremely satisfied.
Time Frame: Day 1
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Decision Aid | No Decision Aid (Control)
Number analyzed (Participants) | 45 | 45
units on a scale | 9.5 (0.13) | 9.4 (0.16)

6. Secondary Outcome: Change in Decision Regret Scale After 6 Weeks and 6 Months
Description: Change in the Decision Regret Scale, which measures distress or remorse after a health care decision. The scale consists of 5 questions, which range from strongly agree to strongly disagree, scoring 0-100 with higher scores indicating more regret.
Time Frame: 6 week and 6 month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Decision Aid | No Decision Aid (Control)
Number analyzed (Participants) | 45 | 45
units on a scale
  Decision regret at 6 weeks | 20 (2.7) | 26 (3.1)
  Decision regret at 6 months | 23 (3.3) | 27 (3.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Decision Aid | No Decision Aid (Control)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/24/NCT03181724/Prot_SAP_000.pdf